CLINICAL TRIAL: NCT05898542
Title: Nature-based Therapies Supporting Conventional Therapies in Promoting Stroke Rehabilitation: a Randomised Controlled Pilot Study.
Brief Title: Nature-based Therapies in Stroke Rehabilitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Joint Authority for Päijät-Häme Social and Health Care (Other)
Collaborators: Helsinki University Central Hospital (Other); University of Jyvaskyla (Other); Tampere University (Other); University of Eastern Finland (Other); Natural Resources Institute Finland (Other Government); University of Helsinki (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Q062
Record Dates: First submitted 2023-06-02; First posted 2023-06-12 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Rehabilitation; Stroke
Keywords: rehabilitation; stroke; nature-based; therapy; microbiome; gut-brain axis
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Randomised controlled study, intervention and control groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nature-based therapy intervention group (Experimental): Patients getting additional therapies outdoors
  Interventions: Procedure: Nature-based therapy
- Control group (No Intervention): Patients getting additional rehabilitation tasks indoors

INTERVENTIONS:
Procedure: Nature-based therapy — Therapy sessions conducted outdoors
  Arms: Nature-based therapy intervention group

SUMMARY:
Stroke rehabilitation patients are subjected to additional nature-based therapies during a rehabilitation ward period.

DETAILED DESCRIPTION:
Inward stroke rehabilitation patients are selected randomly into two groups: intervention and control groups in proportions 1-2:1. Blood samples and microbiome samples of saliva, skin and feces are taken from all patients prior to interventions. These are controlled after 4 weeks from the beginning of the study and 3 months after signing-off the ward. Questionnaires eg on moods, life quality and function deficits are conducted in the beginning of the study, after 4 weeks from the start and 3 months after signing-off. Physiological measurements will be done to observe autonomic nerve status. The interventions consisting of therapy sessions in the hospital nearby nature will be conducted thrice a week one of them being an individual nature-visit with the research worker, one in group and one with family-member or volunteer. The moods and quality of life of the family-member participating in the study will also be followed up. The control group is advised to do simple, more conventional rehabilitative tasks indoors.

ELIGIBILITY:
Inclusion Criteria:

* Acute/Subacute stroke
* Rehabilitation ward patient

Exclusion Criteria:

* Incapable of independent decision making
* Traumatic bleeding in brain tissue
* Severe aphasia
* Severe, malign ongoing disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-31 (Actual); Primary Completion 2026-03-28 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Functional ability | 0-30 days
  Evaluation of functional ability in intervention and control groups by Patient-Reported Outcomes Measurement Information (PROMIS) questionnaire

SECONDARY OUTCOMES:
Quality of life by WHO Disability Assessment Schedule (WHODAS) | 0-30 days
  Evaluation of quality of life in intervention and control groups, measured by WHODAS questionnaire.
Assessment of the intervention impacts on rehabilitation | 0-120 days
  Evaluation of the impact of intervention into achieving the predetermined goals of rehabilitation. Measured by Goal Attainment Scale (GAS) in intervention and control group.
Psychological or psychotherapeutic effects | 0-30 days
  Evaluation of the effect of interventions to psychological well-being or psychotherapeutic effect in comparison to control groups. Measurement by Core-10-survey.
Intervention effects on microbiome | 0-120 days
  Measurement of the effect of intervention on participant microbiome compared to participant microbiome in the control group. Microbial analyses of stool, saliva and flakes of skin.
Intervention effect on the activity of autonomic nerve system | 0-30 days
  The activity of autonomic nerve system is measured with a portable device recording eg heart rate and activity. The activity of autonomic nerve system is measured both in intervention and control group.

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Haveri, MD PhD, Study Director — Päijät-Hämeen Hyvinvointialue
Locations (1):
- Joint Authority for Päijät-Häme Social and Health Care, Lahti, Finland

IPD SHARING:
Plan to Share IPD: No